CLINICAL TRIAL: NCT05357365
Title: A Study on the Establishment of a Cohort for Occupational Disease, Damage Prevention, and Health Management of Emergency Medical Workers
Brief Title: Establishing a Cohort for Occupational Disease of Emergency Medical Workers
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-11-032-003
Record Dates: First submitted 2022-04-03; First posted 2022-05-02 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-06

CONDITIONS: Occupational Diseases; Emergency Departments
MeSH Terms: conditions — Occupational Diseases; Emergencies | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Doctor: Doctors of the Emergency department conduct questionnaires about occupational, mental, physical factors on their health.
  Interventions: Other: questionnaire survey
- Nurses: Nurses of the Emergency department conduct questionnaires about occupational, mental, physical factors on their health.
  Interventions: Other: questionnaire survey

INTERVENTIONS:
Other: questionnaire survey — Questionnaire survey about occupational, mental, physical factors on one's health.

SUMMARY:
This study aims to understand the epidemiological characteristics, related factors , and current status of occupational diseases and damage that occur in emergency medical workers (doctors and nurses). A number of surveys were conducted on about 100 emergency medical workers for about a year with occupational factors, physical health, and mental health.

DETAILED DESCRIPTION:
* Background :

  1. The importance and public role of emergency medical care

     * Emergency medical care is a public and essential medical service that is directly related to the lives of the public and plays a key role in the domestic medical delivery system.
  2. Health problems of domestic emergency medical staff

     * Emergency medical workers are at higher risk than the general population due to higher work intensity, lack of medical staff, unplanned patient occurrence, and congestion.
     * Most emergency medical workers in Korea are classified as high-risk medical staff and receive special medical checkups once or twice a year. On the other hand, these regular medical checkups are only an evaluation of the overall health status of medical staff, which does not lead to prevention before the deterioration of the health status of individual medical staff.
* Objective : The purpose of this study is to establish a cohort research system to develop prevention and health care solutions by identifying epidemiological characteristics, related factors for occupational diseases, and damage occurring in emergency medical workers (doctors and nurses).
* Design: Observational (Cohort study)
* Setting: In the Department of Emergency at the Samsung Medical Center and other hospitals
* Enrollment : About 100 Emergency medical workers (doctors and nurses)
* Methods: Questionnaire surveys on occupational, mental, physical factors during about 1 year.

ELIGIBILITY:
Inclusion criteria: The emergency medical workers

* who have heard the explanation of the study and agreed to participate
* aged 18 or older
* have no occupational disease or damage (within 4 weeks) at the time of cohort establishment.

Exclusion criteria:

* Those who disagree with this study
* A person who is not engaged in actual work, such as taking leave of absence, or who does not agree to participate
* Those with occupational diseases or damage at the time of cohort establishment (within 4 weeks)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Medical workers of the emergency department in the tertiary hospitals in Korea
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Stress_1 | At the enrollment
  Stress of the participants with surveys asking their status
Stress_2 | 3 months after the enrollment
  Stress of the participants with surveys asking their status
Stress_3 | 6 months after the enrollment
  Stress of the participants with surveys asking their status
Stress_4 | 9 months after the enrollment
  Stress of the participants with surveys asking their status
Stress_5 | 12 months after the enrollment
  Stress of the participants with surveys asking their status
Burn out_1 | At the enrollment
  Burn out of the participants with surveys asking their status
Burn out_2 | 3 months after the enrollment
  Burn out of the participants with surveys asking their status
Burn out_3 | 6 months after the enrollment
  Burn out of the participants with surveys asking their status
Burn out_4 | 9 months after the enrollment
  Burn out of the participants with surveys asking their status
Burn out_5 | 12 months after the enrollment
  Burn out of the participants with surveys asking their status
Depression_1 | At the enrollment
  Depression of the participants with surveys asking their status
Depression_2 | 3 months after the enrollment
  Depression of the participants with surveys asking their status
Depression_3 | 6 months after the enrollment
  Depression of the participants with surveys asking their status
Depression_4 | 9 months after the enrollment
  Depression of the participants with surveys asking their status
Depression_5 | 12 months after the enrollment
  Depression of the participants with surveys asking their status
PTSD_1 | At the enrollment
  PTSD of the participants with surveys asking their status
PTSD_2 | 3 months after the enrollment
  PTSD of the participants with surveys asking their status
PTSD_3 | 6 months after the enrollment
  PTSD of the participants with surveys asking their status
PTSD_4 | 9 months after the enrollment
  PTSD of the participants with surveys asking their status
PTSD_5 | 12 months after the enrollment
  PTSD of the participants with surveys asking their status

SECONDARY OUTCOMES:
Circulatory mechanical disease_1 | At the enrollment
  Circulatory mechanical disease of the participants with surveys asking their status
Circulatory mechanical disease_2 | 12 months after the enrollment
  Circulatory mechanical disease of the participants with surveys asking their status
Musculoskeletal disorder_1 | At the enrollment
  Musculoskeletal disorder of the participants with surveys asking their status
Musculoskeletal disorder_2 | 3 months after the enrollment
  Musculoskeletal disorder of the participants with surveys asking their status
Musculoskeletal disorder_3 | 6 months after the enrollment
  Musculoskeletal disorder of the participants with surveys asking their status
Musculoskeletal disorder_4 | 9 months after the enrollment
  Musculoskeletal disorder of the participants with surveys asking their status
Musculoskeletal disorder_5 | 12 months after the enrollment
  Musculoskeletal disorder of the participants with surveys asking their status
Respiratory disease_1 | At the enrollment
  Respiratory disease of the participants with surveys asking their status
Respiratory disease_2 | 12 months after the enrollment
  Respiratory disease of the participants with surveys asking their status
Endocrine/metabolic disease_1 | At the enrollment
  Endocrine/metabolic disease of the participants with surveys asking their status
Endocrine/metabolic disease_2 | 12 months after the enrollment
  Endocrine/metabolic disease of the participants with surveys asking their status
Cancer disease_1 | At the enrollment
  Cancer disease of the participants with surveys asking their status
Cancer disease_2 | 12 months after the enrollment
  Cancer disease of the participants with surveys asking their status
Other diseases_1 | At the enrollment
  Other diseases of the participants with surveys asking their status
Other diseases_2 | 12 months after the enrollment
  Other diseases of the participants with surveys asking their status
The change of how good the participants feel about their health condition (very good~very bad) and checking whether they were sick or feel uncomfortable or not (yes vs. no) | Every 2 weeks from the enrollment up to 1 year
  The change of how good the participants feel about their health condition (very good~very bad) and checking whether they were sick or feel uncomfortable or not (yes vs. no)
Occupational factors of the participants with surveys: Main working hours_1 | At the enrollment
  Main working hours
Occupational factors of the participants with surveys: Main working hours_2 | 1 months after the enrollment
  Main working hours
Occupational factors of the participants with surveys: Main working hours_3 | 2 months after the enrollment
  Main working hours
Occupational factors of the participants with surveys: Main working hours_4 | 3 months after the enrollment
  Main working hours
Occupational factors of the participants with surveys: Main working hours_5 | 4 months after the enrollment
  Main working hours
Occupational factors of the participants with surveys: Main working hours_6 | 5 months after the enrollment
  Main working hours
Occupational factors of the participants with surveys: Main working hours_7 | 6 months after the enrollment
  Main working hours
Occupational factors of the participants with surveys: Main working hours_8 | 7 months after the enrollment
  Main working hours
Occupational factors of the participants with surveys: Main working hours_9 | 8 months after the enrollment
  Main working hours
Occupational factors of the participants with surveys: Main working hours_10 | 9 months after the enrollment
  Main working hours
Occupational factors of the participants with surveys: Main working hours_11 | 10 months after the enrollment
  Main working hours
Occupational factors of the participants with surveys: Main working hours_12 | 11 months after the enrollment
  Main working hours
Occupational factors of the participants with surveys: Main working hours_13 | 12 months after the enrollment
  Main working hours
Occupational factors of the participants with surveys: Average working hours per day_1 | At the enrollment
  Average working hours per day
Occupational factors of the participants with surveys: Average working hours per day_2 | 1 months after the enrollment
  Average working hours per day
Occupational factors of the participants with surveys: Average working hours per day_3 | 2 months after the enrollment
  Average working hours per day
Occupational factors of the participants with surveys: Average working hours per day_4 | 3 months after the enrollment
  Average working hours per day
Occupational factors of the participants with surveys: Average working hours per day_5 | 4 months after the enrollment
  Average working hours per day
Occupational factors of the participants with surveys: Average working hours per day_6 | 5 months after the enrollment
  Average working hours per day
Occupational factors of the participants with surveys: Average working hours per day_7 | 6 months after the enrollment
  Average working hours per day
Occupational factors of the participants with surveys: Average working hours per day_8 | 7 months after the enrollment
  Average working hours per day
Occupational factors of the participants with surveys: Average working hours per day_9 | 8 months after the enrollment
  Average working hours per day
Occupational factors of the participants with surveys: Average working hours per day_10 | 9 months after the enrollment
  Average working hours per day
Occupational factors of the participants with surveys: Average working hours per day_11 | 10 months after the enrollment
  Average working hours per day
Occupational factors of the participants with surveys: Average working hours per day_12 | 11 months after the enrollment
  Average working hours per day
Occupational factors of the participants with surveys: Average working hours per day_13 | 12 months after the enrollment
  Average working hours per day
Occupational factors of the participants with surveys: Damages_1 | At the enrollment
  Damages that occurred while performing business operations
Occupational factors of the participants with surveys: Damages_2 | 3 months after the enrollment
  Damages that occurred while performing business operations
Occupational factors of the participants with surveys: Damages_3 | 6 months after the enrollment
  Damages that occurred while performing business operations
Occupational factors of the participants with surveys: Damages_4 | 9 months after the enrollment
  Damages that occurred while performing business operations
Occupational factors of the participants with surveys: Damages_5 | 12 months after the enrollment
  Damages that occurred while performing business operations
Lifestyle of the participants with surveys: Drinking alcohol status_1 | At the enrollment
  Drinking alcohol status
Lifestyle of the participants with surveys: Drinking alcohol status_2 | 3 months after the enrollment
  Drinking alcohol status
Lifestyle of the participants with surveys: Drinking alcohol status_3 | 6 months after the enrollment
  Drinking alcohol status
Lifestyle of the participants with surveys: Drinking alcohol status_4 | 9 months after the enrollment
  Drinking alcohol status
Lifestyle of the participants with surveys: Drinking alcohol status_5 | 12 months after the enrollment
  Drinking alcohol status
Lifestyle of the participants with surveys : Smoking_1 | At the enrollment
  Smoking status
Lifestyle of the participants with surveys : Smoking_2 | 3 months after the enrollment
  Smoking status
Lifestyle of the participants with surveys : Smoking_3 | 6 months after the enrollment
  Smoking status
Lifestyle of the participants with surveys : Smoking_4 | 9 months up to 1 year
  Smoking status
Lifestyle of the participants with surveys : Smoking_5 | 12 months up to 1 year
  Smoking status
Lifestyle of the participants with surveys : Obesity and weight control_1 | At the enrollment
  Status of obesity and weight control
Lifestyle of the participants with surveys : Obesity and weight control_2 | 3 months after the enrollment
  Status of obesity and weight control
Lifestyle of the participants with surveys : Obesity and weight control_3 | 6 months after the enrollment
  Status of obesity and weight control
Lifestyle of the participants with surveys : Obesity and weight control_4 | 9 months after the enrollment
  Status of obesity and weight control
Lifestyle of the participants with surveys : Obesity and weight control_5 | 12 months after the enrollment
  Status of obesity and weight control
Lifestyle of the participants with surveys: physical activity and exercise_1 | At the enrollment
  Status of physical activity and exercise
Lifestyle of the participants with surveys: physical activity and exercise_2 | 3 months after the enrollment
  Status of physical activity and exercise
Lifestyle of the participants with surveys: physical activity and exercise_3 | 6 months after the enrollment
  Status of physical activity and exercise
Lifestyle of the participants with surveys: physical activity and exercise_4 | 9 months after the enrollment
  Status of physical activity and exercise
Lifestyle of the participants with surveys: physical activity and exercise_5 | 12 months after the enrollment
  Status of physical activity and exercise
Lifestyle of the participants with surveys : A sense of safety_1 | At the enrollment
  A sense of safety
Lifestyle of the participants with surveys : A sense of safety_2 | 3 months after the enrollment
  A sense of safety
Lifestyle of the participants with surveys : A sense of safety_3 | 6 months after the enrollment
  A sense of safety
Lifestyle of the participants with surveys : A sense of safety_4 | 9 months after the enrollment
  A sense of safety
Lifestyle of the participants with surveys : A sense of safety_5 | 12 months after the enrollment
  A sense of safety
Lifestyle of the participants with surveys : Stress level_1 | At the enrollment
  Stress level
Lifestyle of the participants with surveys : Stress level_2 | 3 months after the enrollment
  Stress level
Lifestyle of the participants with surveys : Stress level_3 | 6 months after the enrollment
  Stress level
Lifestyle of the participants with surveys : Stress level_4 | 9 months after the enrollment
  Stress level
Lifestyle of the participants with surveys : Stress level_5 | 12 months after the enrollment
  Stress level
Lifestyle of the participants with surveys: Sleep_1 | At the enrollment
  Sleep
Lifestyle of the participants with surveys: Sleep_2 | 3 months after the enrollment
  Sleep
Lifestyle of the participants with surveys: Sleep_3 | 6 months after the enrollment
  Sleep
Lifestyle of the participants with surveys: Sleep_4 | 9 months after the enrollment
  Sleep
Lifestyle of the participants with surveys: Sleep_5 | 12 months after the enrollment
  Sleep

CONTACTS AND LOCATIONS:
Overall Officials: Taerim Kim, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
This is a multicentered study and there are researchers of other institutes, therefore, IPD can be available to them.